CLINICAL TRIAL: NCT03804957
Title: The Incidence of Pneumothorax After CT-guided Lung Biopsy Performed With and Without Autologous Blood Patching: a Randomized Single-center Prospective Study
Brief Title: Pneumothorax After CT-guided Lung Biopsy: Standard vs Autologous Blood Patching
Acronym: BloodyBiopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICH-BloodyBiopsy
Record Dates: First submitted 2018-12-24; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Pneumothorax; Biopsy Wound
Keywords: biopsy; pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Intervention Model Description: Randomized two arms single center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-guided core needle biopsy (CNB) (Active Comparator): 18 gauge ct-guided lung biopsy
  Interventions: Other: CT-guided core needle biopsy (CNB)
- CNB followed by ABPI. (Experimental): 17 gauge coaxial needle for a 18g ct-guided lung biopsy followed by autologous blood patch injection
  Interventions: Other: Autologous blood patch injection (ABPI)

INTERVENTIONS:
Other: Autologous blood patch injection (ABPI) — Autologous blood patch injection (ABPI) through a coaxial needle at the site of biopsy
  Arms: CNB followed by ABPI.
Other: CT-guided core needle biopsy (CNB) — Standard 18g lung core biopsy
  Arms: CT-guided core needle biopsy (CNB)

SUMMARY:
The aim of this prospective, randomized study is to compare the rate of postoperative pneumothorax between standard CT-guided core needle biopsy (CNB) versus CNB followed by autologous blood patch injection (ABPI).

DETAILED DESCRIPTION:
Pneumothorax is the most common complication of percutaneous lung biopsies. Reducing this risk is a goal of those who perform these procedures, particularly a reduction in large pneumothoraces requiring intervention (eg, pleural drainage) and hospitalization (Clayton et al. 2016). Recently, autologous blood patch injection (ABPI) inside the biopsy track has been suggested as an effective mean of sealing the punctured lung thus halting air loss and consequently pneumothorax (Graffy et al. 2017).

The aim of this prospective, randomized study is to compare the rate of postoperative pneumothorax between standard CT-guided core needle biopsy (CNB) versus CNB followed by ABPI.

In particular, the main objectives are to compare:

1. incidence of immediate pneumothorax
2. incidence of late pneumothorax (2 hrs)
3. incidence of chest tube placement
4. duration of the procedure

ELIGIBILITY:
All patients scheduled for lung biopsy will be asked to join this study. After signing the informed consent the subject will be randomized for ABPI vs CNB approach.

Inclusion criteria:

1) patients with pulmonary nodule requiring CT-guided lung biopsy.

Exclusion criteria:

1. unfit for lung biopsy (INR >1.5, PLT <50.000, single lung);
2. unavailable venous access.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Early Pneumothorax after biopsy | Immediately after lung puncture
  Early Pneumothorax after biopsy as seen by immediate post-biopsy CT and X-ray

SECONDARY OUTCOMES:
Late Pneumothorax after biopsy | 2-6 hours
  Delayed Pneumothorax after biopsy as seen by X-ray after 2-6 hours

CONTACTS AND LOCATIONS:
Overall Officials: EZIO LANZA, MD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- Humanitas Research Hospital, Rozzano, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Maybody M, Muallem N, Brown KT, Moskowitz CS, Hsu M, Zenobi CL, Jihad M, Getrajdman GI, Sofocleous CT, Erinjeri JP, Covey AM, Brody LA, Yarmohammadi H, Deipolyi AR, Bryce Y, Alago W, Siegelbaum RH, Durack JC, Gonzalez-Aguirre AJ, Ziv E, Boas FE, Solomon SB. Autologous Blood Patch Injection versus Hydrogel Plug in CT-guided Lung Biopsy: A Prospective Randomized Trial. Radiology. 2019 Feb;290(2):547-554. doi: 10.1148/radiol.2018181140. Epub 2018 Nov 27. PMID 30480487
- [Result] Graffy P, Loomis SB, Pickhardt PJ, Lubner MG, Kitchin DR, Lee FT Jr, Hinshaw JL. Pulmonary Intraparenchymal Blood Patching Decreases the Rate of Pneumothorax-Related Complications following Percutaneous CT-Guided Needle Biopsy. J Vasc Interv Radiol. 2017 Apr;28(4):608-613.e1. doi: 10.1016/j.jvir.2016.12.1217. Epub 2017 Feb 6. PMID 28185770